CLINICAL TRIAL: NCT04744779
Title: Effectiveness of Office Based Vergence/Accommodative Therapy for the Treatment of Intermittent Exotropia: A Randomized Clinical Trial
Brief Title: Office Based Vergence/Accommodative Therapy for the Treatment of Intermittent Exotropia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sun Yat-sen University (Other)
Collaborators: Salus University (Other)
Responsible Party: Principal Investigator, Ying Kang, Associate Professor of Ophthalmology, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: XT4
Record Dates: First submitted 2021-02-04; First posted 2021-02-09 (Actual); Last update posted 2021-02-23 (Actual); Status verified 2021-02

CONDITIONS: Intermittent Exotropia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Observation (No Intervention): Observation only.
- Office-based accommodative/vergence therapy and home reinforcement (Experimental): Office-based accommodative/vergence therapy (60 minutes per visit, one time per week, 16 weeks) and home reinforcement (15 minutes each time, five times per week, 16 weeks)
  Interventions: Behavioral: Office-based accommodative/vergence therapy and home reinforcement

INTERVENTIONS:
Behavioral: Office-based accommodative/vergence therapy and home reinforcement — Office-based accommodative/vergence therapy (60 minutes per visit, one time per week, 16 weeks) and home reinforcement (15 minutes each time, five times per week, 16 weeks)
  Arms: Office-based accommodative/vergence therapy and home reinforcement

SUMMARY:
Effectiveness of office based vergence/accommodative therapy for the treatment of intermittent exotropia is investigated through a randomized clinical trial

DETAILED DESCRIPTION:
Purpose of study:

i) To evaluate the short-term effectiveness of office based vergence/accommodative therapy (OBVAT) for improving control of intermittent exotropia compared to observation alone; ii) To evaluate the long-term effectiveness of OBVAT for improving control of intermittent exotropia compared to observation alone; iii) To determine the natural history of intermittent exotropia among patients aged 6 to < 18 years who have baseline near stereoacuity of 400 arc sec or better using the Preschool Randot stereotest

ELIGIBILITY:
Inclusion Criteria:

1. 6 to <18 years old
2. Distance exodeviation between 10 and 30 prism diopters (PD) measured by prism and alternate cover test (PACT)
3. Near deviation not exceeding the distance deviation by >10PD by PACT (i.e., convergence insufficiency type intermittent exotropia excluded)
4. Control of deviation meeting all the following criteria based on the office control score scale:

   4.1 Intermittent or constant exotropia at distance (mean of 3 baseline assessments of distance control ≥ Grade 2)# 4.2 Intermittent exotropia or exophoria at near (at least 1 of 3 assessments of near control at the baseline visit Grade 0-4) or orthophoria
5. Stereoacuity: near stereoacuity of 400 arcsec or better by the Preschool Randot stereotest
6. Cycloplegic subjective refraction spherical equivalent (SE) refractive error between -6.00 diopters (D)and +3.50 D inclusive in either eye
7. Must be wearing the updated refractive correction (spectacles) for at least 2 weeks if refractive error (based on cycloplegic subjective refraction performed within 6 months) meets any of the following:

   7.1 Myopia >-0.50 D spherical equivalent in either eye 7.2 Anisometropia >1.00 D spherical equivalent 7.3 Astigmatism in either eye >1.50 D
8. Refractive correction must meet the following guidelines:

   8.1 Anisometropia spherical equivalent must be within 0.25 D of the full anisometropic difference 8.2 Astigmatism cylinder must be within 0.25 D of full correction and axis must be within 5 degree 8.3 For hyperopia and myopia, the spherical component can be reduced by investigator discretion provided reduction is symmetrical and results in residual (i.e., uncorrected) spherical equivalent refractive error that does not exceed +3.50 D spherical equivalent hyperopia or -0.50 D spherical equivalent myopia
9. Gestational age >34 weeks
10. Birth weight >1500 g
11. No previous surgical or nonsurgical treatment for intermittent exotropia other than single vision refractive correction (e.g. progressive addition lens, bifocals, patching, or deliberate over-minus with spectacles >0.50 D)
12. No prior office-based vision therapy for any reason
13. No prior strabismus surgery or botulinum injection, intraocular surgery, or refractive surgery
14. No planned strabismus surgery
15. Visual acuity correctable to at least 20/25 or better at distance and near in each eye.

    * Inclusion criteria 4.1 may be changed to "Intermittent or constant exotropia at distance (mean of 3 baseline assessments of distance control ≥ Grade 1" if there is difficulty in patient recruitment.

Exclusion Criteria:

1. Amblyopia, nystagmus, restrictive or paretic strabismus
2. Regular use of any ocular or systemic medications known to affect accommodation or vergence system, such as atropine, pirenzepine, and anti-epileptic medications, in the most recent 3 months
3. Developmental disability, attention-deficit/hyperactivity disorder (ADHD), or learning disability diagnosis in children that in the investigator's discretion would interfere with office-based treatment
4. Relocation anticipated within 2 year
5. Significant ocular or neurologic disorders (e.g. cerebral palsy) other than strabismus
6. Vertical deviation greater than 3 pd
7. Household member already in the study

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Estimated)
Dates: Start 2021-03 (Estimated); Primary Completion 2023-06 (Estimated); Study Completion 2023-06 (Estimated)

PRIMARY OUTCOMES:
Comparison of the distant office control score between two groups at the primary outcome visit | 16 months
  Comparison of the distant office control score between two groups at the primary outcome visit

SECONDARY OUTCOMES:
Comparison of percentage of patients showing ≥ 1 point change and ≥ 2 points change in office control score | 16 months
  Comparison of percentage of patients showing ≥ 1 point change and ≥ 2 points change in office control score

OTHER OUTCOMES:
Comparison of deterioration rate between 2 groups | 16 months
  Comparison of deterioration rate between 2 groups

IPD SHARING:
Plan to Share IPD: No